CLINICAL TRIAL: NCT06186219
Title: Open-label Study of Rituximab (RTX) Pretreatment Followed by Standard of Care (SOC) Methotrexate-Pegloticase (MTXPEG) to Treat Poorly Controlled Tophaceous Gout in Individuals With Prior Loss of Response to Pegloticase.
Brief Title: Recapturing Immune Tolerance to Pegloticase for the Management of Tophaceous Gout
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, John D. Fitzgerald, MD, PhD, Clin Prof, Clinical Chief, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEG study
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-04

CONDITIONS: Tophaceous Gout
Keywords: gout; pegloticase; rituximab
MeSH Terms: conditions — Gout | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab (Experimental): Rituximab 1000 mg will be administered at week -6 and week -4 via intravenous infusion over the duration of 5 hours prior to the Pegloticase (Standard-of-Care) treatment.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab is a monoclonal antibody that targets cluster of differentiate 20 (CD20) present on B-cells and lowers humoral immunity. Rituximab has been used successfully as a desensitization agent to treat Highly Human Leukocyte Antigens (HLA)-sensitized patients planning renal transplant. All cases of antibody-mediated rejection were seen in the placebo group, none in the Rituximab group. Rituximab has been safely used with Methotrexate in the treatment of Rheumatoid Arthritis, where co-administration of Methotrexate and Rituximab results in better outcomes than either medication alone.
  We propose this safety and feasibility open-label trial that will examine if Rituximab pre-treatment before Standard-of-Care Methotrexate-Pegloticase will result in recapture of Pegloticase efficacy as measured by serum urate (SU) < 6 mg/dL throughout the trial and up to 6-months of Methotrexate-Pegloticase administration.

SUMMARY:
This safety and feasibility, open-label study of up to 9 subjects will examine a group of subjects with poorly controlled tophaceous gout (intolerant to or ineffective oral urate lowering agents and loss of prior Pegloticase response) pre-treated with Rituximab to recapture response to Methotrexate-Pegloticase.

DETAILED DESCRIPTION:
Rituximab 1000 mg will be administered at week -6 and week -4 via intravenous infusion over the duration of 5 hours prior to Methotrexate-Pegloticase Standard-of-Care treatment. Per FDA approved dosing in the package insert, Rituximab infusion with concentration of 10 mg/mL will begin at 50 mg/hr. In the absence of infusion toxicity, increase infusion rate by 50 mg/hour increments every 30 minutes, to a maximum of 400 mg/hour or total dose of 1000 mg.

All subjects will be treated with Methotrexate-Pegloticase Standard-of-Care with FDA-approved dosing of Pegloticase 8 mg IV infusion every 2 weeks, co-administered with methotrexate 15 mg orally once weekly (started 4 weeks prior to Pegloticase initiation).

Standard-of-Care includes Pegloticase infusion every 2 weeks as long as clinically indicated (e.g., persistent tophus), concluding treatment when all tophaceous gout lesions resolve or up to 12-months, safety stop point, or subject withdrawal from the study.

Subjects will be on study for up to 24 months. Screening visit: up to 28-days.

Treatment visit:

1. Rituximab Pre-Treatment: up to 6-weeks + 1 week prior to Pegloticase treatment. (Pre-treatment of Rituximab will occur at -6 and -4 weeks.)
2. Methotrexate Treatment (Standard-of-Care): up to 6 weeks + 1 week prior to Pegloticase treatment. (Administered four weeks prior to Pegloticase and weekly during Pegloticase treatment).
3. Methotrexate-Pegloticase Study Treatment (Standard-of-Care): up to 12 months of Standard-of-Care. (Methotrexate is administered weekly and Pegloticase is coadministered every two weeks).

Follow-up phone visits: up to 30 and 60 days after last dose of Methotrexate-Pegloticase + 7 days.

Total subject participation duration is up to 24 months. Total study duration for recruitment, enrollment, and study completion of all subjects is up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet/provide all the following criteria:

1. Must be able to provide written informed consent.
2. Male or female ≥ 18 years of age at Baseline Visit.
3. Meets the American College of Rheumatology Classification Criteria for Gout.
4. Poorly controlled tophaceous gout, defined as meeting the following criteria:

   1. Hyperuricemia during the screening period defined as serum urate ≥ 6 mg/dL.
   2. Failure to maintain normalization of serum urate with xanthine oxidase inhibitors at the maximum medically appropriate dose, or with a contraindication to xanthine oxidase inhibitor therapy based on medical record review or subject interview, and;
   3. Symptoms of gout including at least 1 of the following:

   i. Presence of at least one tophus. ii. Recurrent flares defined as 2 or more flares in the past 12 months prior to screening.
5. Prior discontinued use of Pegloticase due to failure (rising SU > 6 mg/dL or history of moderate to severe infusion reaction).
6. Normal Glucose-6-phosphate dehydrogenase levels.
7. Willing to discontinue any oral urate lowering therapy for at least 7 days prior to first Pegloticase infusion and remain off therapy when receiving Pegloticase infusions.
8. Women of childbearing potential (including those with an onset of menopause <2 years prior to screening, non-therapy-induced amenorrhea for <12 months prior to screening, or not surgically sterile [absence of ovaries and/or uterus]) must have negative serum/urine pregnancy tests during Screening and Week 0; subjects must agree to use reliable form of contraception during the study. Hormonal contraception must be continued while on Methotrexate. Highly effective contraceptive methods (with a failure rate <1% per year), when used consistently and correctly, include implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence, or vasectomized partner.

Exclusion Criteria:

Subjects will be ineligible for trial participation if they meet any of the following criteria:

1. Glucose-6-phosphate dehydrogenase deficiency (documented or tested at the Screening Visit).
2. Chronic renal impairment defined as estimated glomerular filtration rate (epidermal growth factor receptor) < 30 mL/min/1.73 m2 or currently on dialysis.
3. Non-compensated congestive heart failure (stage C) or hospitalization for congestive heart failure within 3 months of the Screening Visit, uncontrolled arrhythmia.
4. Treatment for acute coronary syndrome (myocardial infarction or unstable angina).
5. Uncontrolled blood pressure (>160/100 mmHg) prior to Rituximab infusion (week -6, week -4).
6. On treatment for current non-skin cell cancer.
7. Any serious acute bacterial infection, unless treated and completely resolved with antibiotics at least 2 weeks prior to the Week -6 Visit.
8. Severe chronic or recurrent bacterial infections, such as recurrent pneumonia or chronic bronchiectasis.
9. Anaphylaxis or other prior severe infusion reaction to Pegloticase that the study allergy-immunologist deems treatment with Pegloticase to be unsafe to rechallenge.
10. History of any transplant surgery requiring maintenance immunosuppressive therapy.
11. Known history of hepatitis B virus surface antigen positivity or hepatitis B DNA positivity.
12. Known history of hepatitis C virus ribonucleic acid (RNA) positivity.
13. Known history of Human Immunodeficiency Virus (HIV) positivity.
14. Pregnant, planning to become pregnant, breastfeeding, or not on an effective form of birth control, as determined by the Investigator.
15. Contraindication to Methotrexate treatment or Methotrexate treatment considered inappropriate.
16. Known intolerance to steroids, such as:

    1. History of steroid-induced Psychosis.
    2. History or steroid-induced diabetic ketoacidosis or hyperosmolar.
17. Receipt of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, prior to Methotrexate administration at Week -6 or plans to take an investigational drug during the study.
18. Liver transaminase levels (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) > twice upper limit of normal (ULN) at the Screening Visit).
19. Chronic liver disease.
20. White blood cell count < 3,500/µL, hematocrit < 28 percent, or platelet count < 75,000/µL.
21. Currently receiving systemic or radiologic treatment for ongoing cancer.
22. History of malignancy within 5 years other than non-melanoma skin cancer or in situ carcinoma of cervix.
23. Unsuitable candidate for the study, based on the opinion of the Investigator (e.g., cognitive impairment), such that participation might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or complete the study.
24. Alcohol use in excess of 1 alcoholic beverages per day.
25. Current pulmonary fibrosis, bronchiectasis, or interstitial pneumonitis. If deemed necessary by the Investigator, a chest X-ray may be performed during Screening.
26. Prior treatment with Rituximab (within 6 months) or Methotrexate (within 3 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-04-10 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
The study will be measured by the frequency and grade of adverse event (AEs) (solicited and unsolicited), serious adverse experience (SAEs), adverse event of special interest (AESI1s), medically attended adverse events (MAAEs). | 2 years
  Simple descriptive statistics will be used to summarize toxicities in terms of type, severity and minimum or maximum values for laboratory measures, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects. Safety Analyses will be performed on Safety Analysis Set.
  After the first Pegloticase infusion, any subsequent pre-Pegloticase infusion lab result of serum urate > 6 mg/dL will terminate the study.
Neutralizing antibody titers (assays provided by Horizon labs) will be measured at Screening (Visit 0), prior to first Pegloticase infusion (Visit 3, Week 0), Visit 9, Week 12 and Visit 16, Week 26. | 2 years
  Mean change between baseline and the specified follow up measurements will be analyzed using general linear modelling with adjustment to control for within person correlation of repeated measurements.

CONTACTS AND LOCATIONS:
Overall Officials: John FitzGerald, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No